CLINICAL TRIAL: NCT06994988
Title: Multi-modal Smart Band-Aid for AI-based Quantification of Pain
Brief Title: ARPA-H Smart Band-Aid to Measure Chronic Pain in Women
Status: Not yet recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Tufts University (Other); The Advanced Research Projects Agency for Health (ARPA-H) (Unknown); Walter Reed National Military Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Steven Cohen, Edmond I Eger Professor of Anesthesiology and Vice Chair of Pain Medicine, Northwestern University
Other Study IDs: STU00223452; FP00008853 (Other Grant/Funding Number: Advanced Research Projects Agency for Health)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Smart Band-Aid; A-Band; Chronic Pain; ARPA-H; AI and Chronic Pain; Objective measure; Biomarker
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Chronic pain patients: 85 female patients with chronic pain > 3 months duration
  Interventions: Device: A-Band (Smart Band-Aid); Combination Product: Empatica Smartwatch; Behavioral: Questionnaires: Hospital Anxiety & Depression Scale, Central Sensitization Inventory, Pain Catastrophizing Scale, Somatic Symptom Scale-8, Pain Self-Efficacy Questionnaire-10, Athens Insomnia Scale
- Healthy control patients: 35 healthy control patients
  Interventions: Device: A-Band (Smart Band-Aid); Combination Product: Empatica Smartwatch; Behavioral: Questionnaires: Hospital Anxiety & Depression Scale, Central Sensitization Inventory, Pain Catastrophizing Scale, Somatic Symptom Scale-8, Pain Self-Efficacy Questionnaire-10, Athens Insomnia Scale

INTERVENTIONS:
Device: A-Band (Smart Band-Aid) — The A-Band is a smart band-aid placed on the forearm or other designated site that collects interstitial fluid (ISF) from participants using a microneedle patch. ISF is a natural fluid found between your cells that can inform us on your bodily readings and health. A microneedle patch is a safe alternative to standard fluid collection which uses tiny needles to collect the ISF. The patches consist of single-use, sterile (clean) microneedles created from biocompatible materials. These microneedles penetrate the outermost skin layer without causing significant discomfort, pain, or bleeding.
Combination Product: Empatica Smartwatch — A commercial smart band will be worn by participants for 22+ hours a day for approximately 7 days. The smart band collects biophysical data from the participant. This includes data on biomarkers, heart rate and heart rate variability, galvanic skin response, step count, and temperature fluctuations, among other biophysical data.
Behavioral: Questionnaires: Hospital Anxiety & Depression Scale, Central Sensitization Inventory, Pain Catastrophizing Scale, Somatic Symptom Scale-8, Pain Self-Efficacy Questionnaire-10, Athens Insomnia Scale — HADS- measures anxiety and depression (0-21, higher scores signify greater pathology); CSI- measures central sensitization (0-100, higher scores signify greater central sensitization, PCS- measures catastrophizing (0-52, higher scores signify greater catastrophization), SSS-8- measures somatization (0-32, higher scores signify greater somatization), PSEQ-10- measures self-efficacy (0-60, with lower scores signifying low self-efficacy), AIS- measures sleep (0-28, with higher scores signifying greater sleep dysfunction)

SUMMARY:
The goal of this clinical trial is to test whether a minimally invasive microneedle patch, called the A-Band (Smart Band-aid), worn on the arm (monitoring key biomarkers in interstitial fluid) and a commercial smartwatch can accurately correlate with self-reported pain in women with chronic pain. A secondary purpose of the study is to identify demographic and clinical variables impacting pain measurement.

The main questions that this study aims to answer are:

* What is the correlation between AI-adjusted pain scores, based on biomarkers and validated tools, and self-reported pain scores?
* What influence do demographic and clinical information have in the correlation of these pain scores?

Researchers will compare data from these tools with self-reported pain scores in women with chronic pain and healthy women.

Participants will:

* Be a part of the study for approximately 8 days
* Attend 2-3 in-person visits at the applicable clinical center over approximately one week
* Wear a Smart Band-Aid (A-Band) at least twice per day for a week, with each application lasting up to 90 minutes
* Complete questionnaires regarding medical history, pain information, mental health, sleep, and demographic data
* Record daily pain scores
* Wear a smartwatch for one week which will collect biophysical data (heart rate, skin response, etc.)
* Collect daily saliva samples
* Have blood drawn by medical staff at 2 in-person visits

DETAILED DESCRIPTION:
This study proposes the collection of interstitial fluid (ISF) from participants using a microneedle patch. ISF is a natural fluid found between your cells that can inform us on your bodily readings and health. A microneedle patch is a safe alternative to standard fluid collection which uses tiny needles to collect the ISF. The patches consist of single-use, sterile (clean) microneedles created from biocompatible materials. These microneedles penetrate the outermost skin layer without causing significant discomfort, pain, or bleeding.

The A-Band is an investigational device and has not been approved for use by the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

For chronic pain group:

* Female, 18 years or older.
* Diagnosis of chronic pain condition (e.g., fibromyalgia, chronic lower back pain) as determined by the Principal Investigator.
* Ability to provide informed consent.

For healthy controls:

* Female, 18 years or older.
* No history of chronic pain.
* No significant or poorly controlled medical conditions as determined by the Principal Investigator and exclusion criteria.
* No significant active, poorly controlled psychological conditions as determined by the Principal Investigator and exclusion criteria.
* Ability to provide informed consent.

Exclusion Criteria (both groups):

* Pregnant or breastfeeding women.

  * Substance abuse or psychiatric disorders that interfere with study participation.
  * Major medical conditions (such as severe cardiovascular, neurological, cancer or autoimmune diseases) or psychological conditions (e.g., active, poorly-controlled depression, anxiety disorder, PTSD, substance use disorder) that interfere with study participation.
  * Possibility of secondary financial gain from participation
  * Interventional pain treatment(s) within 6 weeks of baseline (injection, epidural, etc.)
  * Current opioid usage or usage within 2 weeks of baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Biological females with chronic pain and biological females without chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-10-23 (Estimated); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Difference between patient-reported pain score and objective pain score as calculated by AI | Days 0 thru 7, for 8 total days
  We will measure the difference between the patient-reported pain scores and AI-generated objective pain score in subgroups of chronic pain patients (e.g., nociplastic pain, neuropathic pain, nociceptive pain, mixed pain) and healthy controls (if they have acute pain).

SECONDARY OUTCOMES:
Pain Scores from Biochemical and Biophysical Measurements & Instruments Measured from Questionnaires (affective-motivational and cognitive components) | From Day 0 thru Day 7, for 8 total days
  Biomarker readings from interstitial fluid, blood serum, and a commercial smart band will be inserted into an AI machine learning algorithm and combined with the scores on the instruments measuring the affective and cognitive pain components to develop an "objective" pain score. The affective-motivational component will be determined by scores on the Hospital Anxiety & Depression Scale, Somatic Symptom Scale-8 & Athens Insomnia Scale. The cognitive-evaluative component will be determined by scores on the Pain Catastrophizing Scale, Pain Self-Efficacy Questionnaire-10 and Somatic Symptom Scale-8.
Patient-reported pain score | Days 0 thru 7, for 8 total days
  Patient-reported pain scale on a 0-10 pain scale (Defense and Veterans Pain Rating Scale), recorded at least twice per day upon patch application.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request with IRB approval.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: For 3 years after completion of the study
Access Criteria: Investigators with an IRB-approved protocol, after approval from sponsor.

REFERENCES:
- [Background] Guo LL, Pfohl SR, Fries J, Johnson AEW, Posada J, Aftandilian C, Shah N, Sung L. Evaluation of domain generalization and adaptation on improving model robustness to temporal dataset shift in clinical medicine. Sci Rep. 2022 Feb 17;12(1):2726. doi: 10.1038/s41598-022-06484-1. PMID 35177653
- [Background] Wu Z, Yao H, Liebovitz D, Sun J. An iterative self-learning framework for medical domain generalization. Advances in Neural Information Processing Systems. 2024 Feb 13;36.
- [Background] Strawbridge R, Young AH, Cleare AJ. Biomarkers for depression: recent insights, current challenges and future prospects. Neuropsychiatr Dis Treat. 2017 May 10;13:1245-1262. doi: 10.2147/NDT.S114542. eCollection 2017. PMID 28546750
- [Background] Yang J, Luo R, Yang L, Wang X, Huang Y. Microneedle-Integrated Sensors for Extraction of Skin Interstitial Fluid and Metabolic Analysis. Int J Mol Sci. 2023 Jun 8;24(12):9882. doi: 10.3390/ijms24129882. PMID 37373027
- [Background] Diaz MM, Caylor J, Strigo I, Lerman I, Henry B, Lopez E, Wallace MS, Ellis RJ, Simmons AN, Keltner JR. Toward Composite Pain Biomarkers of Neuropathic Pain-Focus on Peripheral Neuropathic Pain. Front Pain Res (Lausanne). 2022 May 11;3:869215. doi: 10.3389/fpain.2022.869215. eCollection 2022. PMID 35634449
- [Background] Telli H, Ozdemir C. Is nociplastic pain, a new pain category, associated with biochemical, hematological, and inflammatory parameters? Curr Med Res Opin. 2024 Mar;40(3):469-481. doi: 10.1080/03007995.2024.2304106. Epub 2024 Jan 22. PMID 38204412
- [Background] Eldabe S, Obara I, Panwar C, Caraway D. Biomarkers for Chronic Pain: Significance and Summary of Recent Advances. Pain Res Manag. 2022 Nov 7;2022:1940906. doi: 10.1155/2022/1940906. eCollection 2022. PMID 36385904
- [Background] Tracey I, Woolf CJ, Andrews NA. Composite Pain Biomarker Signatures for Objective Assessment and Effective Treatment. Neuron. 2019 Mar 6;101(5):783-800. doi: 10.1016/j.neuron.2019.02.019. PMID 30844399